CLINICAL TRIAL: NCT00512512
Title: Transoral Endoscopic Liver Biopsy During Laparoscopic Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Michael Schweitzer, M.D., Johns Hopkins
Other Study IDs: NA_00007226
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2009-07

CONDITIONS: Steatohepatitis; Morbid Obesity
Keywords: transoral; transluminal; endoscopic; laparoscopic; liver; biopsy
MeSH Terms: conditions — Fatty Liver; Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Transoral Endoscopic Liver Biopsy — Liver will be biopsied with transoral endoscope instead of the laparoscopic instruments during laparoscopic gastric bypass

SUMMARY:
This research is being done to evaluate the ability to obtain a liver sample using upper endoscopy rather than through a laparoscopic procedure. The investigators hypothesize that the endoscopic transoral route is as effective as the laparoscopic route.

ELIGIBILITY:
Inclusion Criteria:

1. Any patient who meets criteria to undergo laparoscopic Roux-en Y Gastric Bypass (BMI>40 or BMI>35 with multiple medical co morbidities).
2. Age greater than 18 years.
3. Ability to complete all necessary components of study (gastric bypass surgery standard qualifications).

Exclusion Criteria:

1. Inability to give informed consent
2. Women who are pregnant or in whom pregnancy status cannot be confirmed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Morbid Obese patients who are already approved for gastric bypass surgery.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Schweitzer, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Result] Steele K, Schweitzer MA, Lyn-Sue J, Kantsevoy SV. Flexible transgastric peritoneoscopy and liver biopsy: a feasibility study in human beings (with videos). Gastrointest Endosc. 2008 Jul;68(1):61-6. doi: 10.1016/j.gie.2007.09.040. Epub 2008 Mar 4. PMID 18308313